CLINICAL TRIAL: NCT07273942
Title: Remote Ischemic Postconditioning in Septic Shock
Acronym: RIPOST-sepsis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL24_0937
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Adult Patients With Septic Shock Admitted in Intensive Care Unit
Keywords: Septic shock; Remote conditioning; Ischemic conditioning; Ischemia-reperfusion; Intensive care unit
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Masking Description: In the control group, no intervention is performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic conditioning (Experimental): A brachial cuff is positioned around one arm of the patient. Remote ischemic conditioning consists of alternating inflations and deflations of the brachial cuff. Four cycles of ischemic conditioning (5-min brachial cuff inflation at 200 mmHg followed by 5-min cuff deflation) are started as soon as possible after inclusion. The intervention is repeated 12 and 24 hours after inclusion.
  Interventions: Other: Remote ischemic conditioning
- Control group (Other): No intervention wil be performed in the control group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Remote ischemic conditioning — A brachial cuff is positioned around one arm of the patient. Remote ischemic conditioning consists of alternating inflations and deflations of the brachial cuff. Four cycles of ischemic conditioning (5-min brachial cuff inflation at 200 mmHg followed by 5-min cuff deflation) are started as soon as possible after inclusion. The intervention is repeated 12 and 24 hours after inclusion.
  Arms: Remote ischemic conditioning
Other: No intervention — No intervention will be performed in the conrol group
  Arms: Control group

SUMMARY:
Septic shock is a leading cause of death worldwide despite intensive research efforts. Only a few interventions have been proven to be effective in improving patient-centered outcomes. Recent clinical trials have reported the safety and efficacy of remote ischemic postconditioning (RIPOST) in a variety of pathologies, including myocardial infarction, cardiac surgery, and stroke. While RIPOST was mainly tested in pathologies with low mortality rates, several follow-up studies of large randomized clinical trials in acute myocardial infarction and in patients undergoing coronary artery bypass surgery have reported significant decreases (> 50%) in long-term mortality. Experimental studies and proof-of-concept clinical trials have also suggested the potential benefits of RIPOST on mortality in sepsis and septic shock. The present protocol aims to test whether this non-invasive, widely available, inexpensive, and innovative intervention can improve survival in septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized in intensive care unit for less than 24 hours
* Septic shock (Sepsis-3 definition) evolving for less than 18 hours
* Preliminary written informed consent obtained from the patient or his/her close relative, or use of the emergency procedure in accordance with local regulations

Exclusion Criteria:

* Contraindication of the use of a brachial pressure cuff on both arms
* Cardiac arrest
* Pregnancy or breast feeding
* Participation in another interventional study
* Lack of French national health insurance coverage
* Patient with any legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at day 90 after inclusion | 90 days after inclusion

SECONDARY OUTCOMES:
Functional recovery | Day 90
  Number of days alive after discharge at home by day 90
SF-36 (Short Form-36 Health Survey) questionnaire score | Day 90
  Quality of livre is evaluated by SF-36 (Short Form-36 Health Survey) questionnaire at day 90
Number of days alive without vasopressors | Day 7
Sepsis-related Organ Failure Assessment (SOFA) score | Inclusion and days 1, 3 and 7
  The severity of multiple organ failure assessed by the Sepsis-related Organ Failure Assessment (SOFA) score
Sepsis-induced immuno-inflammatory responses | Inclusion and days 1, 3 and 7
  Dosage of inflammation biomarkers
  * Neutrophils to lymphocytes ratio for all patients
  * In about 100 patients (from two centers) with a biological collection, markers of inflammatory/immune response (including cytokines, monocyte HLA-DR (Human Leukocyte Antigen) expression, immature neutrophils)

CONTACTS AND LOCATIONS:
Locations (23):
- France (23):
  - Service de Réanimation Médicale, Hôpital Jean-Minjoz, CHU de Besançon, Besançon
  - Service Réanimation Polyvalente, Centre Hospitalier de Fleyriat, Bourg-en-Bresse
  - Service de Médecine Intensive- Réanimation, Hôpital Gabriel Montpied, CHU de Clermont-Ferrand, Clermont-Ferrand
  - Service de Médecine Intensive-Réanimation, Hôpital Henri Mondor, Assistance Publique des Hôpitaux de Paris, Créteil
  - Service de Médecine intensive-Réanimation,Hôpital F Mitterrand, CHU de Dijon, Dijon
  - Service de Médecine intensive-Réanimation,Hôpital Albert Michallon, CHU de Grenoble, La Tronche
  - Service de Médecine Intensive-Réanimation, Hôpital Bicêtre, Assistance Publique des Hôpitaux de Paris, Le Kremlin-Bicêtre
  - Service de Médecine Intensive-Réanimation, Hôpital Salengro, CHU de Lille, Lille
  - Service de Médecine Intensive-Réanimation, Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon
  - Service Réanimation Polyvalente, Hôpital Saint-Joseph Saint-Luc, Lyon
  - Service de Médecine Intensive-Réanimation, Hôpital Nord, Assistance Publique des Hôpitaux de Marseille, Marseille
  - Service de Réanimation des Urgences, Hôpital de la Timone, CHU de Marseille, Marseille
  - Service de Médecine intensive-Réanimation, Hôpital Lapeyronie, CHU de Montpellier, Montpellier
  - Service de Médecine Intensive-Réanimation, Hôpital Central, CHRU de Nancy, Nancy
  - Service de Médecine Intensive-Réanimation, Hôtel Dieu, CHU de Nantes, Nantes
  - Service de Médecine Intensive - Réanimation, Hôpital Cochin, Assistance Publique des Hôpitaux de Paris, Paris
  - Service d'Anesthésie - Réanimation - Médecine Intensive, Hôpital Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite
  - Service de Médecine Intensive et Réanimation Polyvalente, Hôpital Robert Debré, CHU Reims, Reims
  - Service des maladies infectieuses et réanimation médicale, Hôpital Pontchaillou, CHU de Rennes, Rennes
  - Service Réanimation Polyvalente, Centre Hospitalier de Roanne, Roanne
  - Service de Médecine intensive-Réanimation, Hôpital Nord, CHU de St Etienne, Saint-Priest-en-Jarez
  - Service de Médecine Intensive-Réanimation, Nouvel Hôpital Civil, CHU de Strasbourg, Strasbourg
  - Service de Médecine Intensive-Réanimation, Hôpital Bretonneau, CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No